CLINICAL TRIAL: NCT04490980
Title: The Analgesic Effect of Butorphanol After Cesarean Section
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tongji Hospital (Other)
Responsible Party: Principal Investigator, Deng Dongrui, professor,chief doctor, Tongji Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TJ-C20200119
Record Dates: First submitted 2020-02-03; First posted 2020-07-29 (Actual); Last update posted 2020-07-29 (Actual); Status verified 2020-06

CONDITIONS: Analgesia
MeSH Terms: conditions — Agnosia | interventions — Butorphanol

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Observed group (Experimental)
  Interventions: Drug: butorphanol
- Control group (No Intervention)

INTERVENTIONS:
Drug: butorphanol — Observed group:Intravenous drip of Butorphanol in patients after cesarean section;control group: intravenous drip of saline in patients after cesarean section
  Arms: Observed group

SUMMARY:
We evaluated the clinical effect of Butorphanol on postoperative analgesia by observing the vital signs of patients, general condition of newborns and pain assessment.

ELIGIBILITY:
Inclusion Criteria:

Healthy women at term (37 to 42 weeks of gestation), who desired cesarean section were eligible to participate. undergoing ；No drug sensitive history

Exclusion Criteria:

Patients with a history of anesthetics allergy and patients with preterm labor, multiple pregnancies and severe obstetric complications

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-08-01 (Estimated); Primary Completion 2020-11-30 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
change from Visual Analogue Score for pain | assess VAS at 24 hours, 25 hours, 26 hours, 27 hours, 30 hours, 36 hours after the cesarean section
  VAS is the most common pain scale for quantification. The score is higher, the patient will be more painful. That will indicate if the analgesia is effective. Visual analog scale (VAS) ranging from 0 to 10 (with 10 representing the worst pain imaginable) to measure the degree of pain for participants

SECONDARY OUTCOMES:
heart rates | at 24 hours, 30 hours, 36 hours after the cesarean section
  heart rates（bpm)
jaundice index of the newborn,1 minute and 5 minutes Apgar score | jaundice index: 24 hours, 48 hours, 72 hours after the cesarean section
  Neonatal Apgar scores at the first and fifth minute.The score indicates the infant s' conditions, including heart rate, breathing, muscle tone, reflex response, color. Each characteristic is given an individual score; two points for each of the five categories if all is completely well; then all scores are totaled. The score is from 0 to 10.
blood pressure | at 24 hours, 30 hours, 36 hours after the cesarean section
  blood pressure(mmHg)
breath | at 24 hours, 30 hours, 36 hours after the cesarean section
  breath(bpm)
pulse | at 24 hours, 30 hours, 36 hours after the cesarean section
  pulse(bpm)

CONTACTS AND LOCATIONS:
Overall Officials: Xun Gong, Study Chair — Tongji Hospital

IPD SHARING:
Plan to Share IPD: No